CLINICAL TRIAL: NCT03134469
Title: Efficacy of Probiotics on Excessive Gas Accumulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Probi AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ProGastro 17
Record Dates: First submitted 2017-04-26; First posted 2017-05-01 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Flatulence; Bloating
MeSH Terms: conditions — Flatulence

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics (Experimental): Intake of a probiotic capsule once daily
  Interventions: Dietary Supplement: Probiotic supplement
- Placebo (Placebo Comparator): Intake of a placebo capsule once daily
  Interventions: Dietary Supplement: Placebo supplement

INTERVENTIONS:
Dietary Supplement: Probiotic supplement — Probiotic supplement
  Arms: Probiotics
Dietary Supplement: Placebo supplement — Placebo supplement
  Arms: Placebo

SUMMARY:
Efficacy of probiotics on excessive gas accumulation

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults 18-50 years, at the time of signing the informed consent.
* Willing and able to give written informed consent for participating in the study
* Willing to comply with all study procedures

Exclusion Criteria:

* Chronic intestinal disease, immunodeficiency disorder or immunosuppressive treatment
* Clinically significant frequent constipation or diarrhea at the screening visit as judged by the Investigator
* Known gluten intolerance, lactose intolerance, milk protein allergy
* Vegetarian diet
* Intake of antibiotics within four weeks prior to the start of the study
* Hypersensitivity to any of the ingredients in the investigational product (IP)
* Regular intake of probiotics within four weeks prior to the start of the study
* History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk if participating in the study, or influence the results or the subject´s ability to participate in the study
* Investigator considers the subject unlikely to comply with study procedures, restrictions and requirements.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2017-04-18 (Actual); Primary Completion 2017-10-19 (Actual); Study Completion 2017-10-19 (Actual)

PRIMARY OUTCOMES:
Breath hydrogen | 4 hours
  The level of breath hydrogen is measured after a challenge with lactulose

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Lund University, Lund
  - CTC Clinical Consultants, Uppsala

IPD SHARING:
Plan to Share IPD: No